CLINICAL TRIAL: NCT00123929
Title: Patterns of Genetic Expression Associated to Sensibility to Doxorubicin Versus Docetaxel as Neoadjuvant Chemotherapy for Locally Advanced Breast Cancer
Brief Title: Genetic Expression and Prediction of Response to Neoadjuvant Docetaxel or Doxorubicin in Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Miguel Martin, MD, Hospital San Carlos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/117
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant chemotherapy; genetic signature; doxorubicin; docetaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): doxorubicin
  Interventions: Drug: doxorubicin
- 2 (Other): docetaxel
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: docetaxel — 100 mg/m2 every 3 weeks times 4
  Other Names: taxotere
  Arms: 2
Drug: doxorubicin — 75 mg/m2 every 3 weeks times 4
  Other Names: adriamycin
  Arms: 1

SUMMARY:
After a core biopsy of the tumor is obtained, patients with locally advanced breast cancer are randomized to receive 4 cycles of full dose doxorubicin (75 mg/m2 e3w) or docetaxel (100 mg/m2 e3w). After the fourth cycle, patients are submitted to surgery to ascertain pathological response. They then receive the opposite drug, hormones, Herceptin, and radiation as indicated.

DETAILED DESCRIPTION:
The aim of the study is to define the genetic signature which predicts the response to single drug doxorubicin versus docetaxel. 250 patients will be included. cDNA microarrays will be produced and the genetic pattern will be correlated with the response to doxorubicin and docetaxel. Secondary aim is the prediction of response by means of IHC determinations (her2, ER, PgR, Ki67, protein TAU), FISH (topoisomerase II alpha, her2) and PCR (topoisomerase II alpha).

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, inoperable breast carcinoma or stage II not amenable to breast preserving surgery (amendment introduced on november 2006)
* Signed informed consent

Exclusion Criteria:

* Age >75
* Cardiac disease; LEFT <50%
* Hyperbilirubinemia

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
correlation of genetic tumoral pattern with response to docetaxel versus doxorubicin | 2005-2009

SECONDARY OUTCOMES:
response rate to doxorubicin versus docetaxel | 2005-2013

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Diaz-Rubio, MD, PhD, Study Director — Servicio de Oncologia Medica, Hospital Universitario San Carlos, Madrid, Spain; Martin Miguel, MD, PhD, Principal Investigator — Hospital San Carlos, Madrid, Spain
Locations (1):
- Servicio de Oncologia Medica, Hospital Clinico San Carlos, Madrid, Spain

REFERENCES:
- [Derived] Ruiz-Pinto S, Martin M, Pita G, Caronia D, de la Torre-Montero JC, Moreno LT, Moreno F, Garcia-Saenz JA, Benitez J, Gonzalez-Neira A. Pharmacogenetic variants and response to neoadjuvant single-agent doxorubicin or docetaxel: a study in locally advanced breast cancer patients participating in the NCT00123929 phase 2 randomized trial. Pharmacogenet Genomics. 2018 Nov;28(11):245-250. doi: 10.1097/FPC.0000000000000354. PMID 30334909